CLINICAL TRIAL: NCT02506816
Title: A Preoperative "Window-opportunity", Multicenter, Pharmacokinetic-pharmacodynamic Study to Evaluate the Inhibitory Effects of Single Agent AZD2281 (Olaparib), in Patients With Early-stage Endometrial Carcinoma
Brief Title: Preoperative Olaparib Endometrial Carcinoma Study (POLEN)
Acronym: Polen
Status: Completed | Type: Observational
Sponsor: MedSIR (Other)
Collaborators: AstraZeneca (Industry); Experior (Industry)
Responsible Party: Sponsor
Other Study IDs: MedOPP044; 2015-001156-30 (EudraCT Number)
Record Dates: First submitted 2015-06-29; First posted 2015-07-23 (Estimated); Results first posted 2019-11-15 (Actual); Last update posted 2020-11-30 (Actual); Status verified 2019-11

CONDITIONS: Endometrial Carcinoma
MeSH Terms: conditions — Endometrial Neoplasms | interventions — olaparib

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Tumor cells Plasma
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Olaparib: Drug exposure has a limited duration 28 (+/- 5) days.
  Interventions: Drug: Olaparib

INTERVENTIONS:
Drug: Olaparib — Drug exposure has a limited duration 28 (+/- 5) days and at lower dose (600mg/day) than therapeutical accepted (800mg/day).
  Other Names: Lynparza

SUMMARY:
The primary objective of this study is to identify, in human tumour samples, biomarker changes associated to short exposure to AZD2281 as potential predictors of activity in Endometrial Carcinoma (EC).

This is an exploratory study with a biological primary endpoint. Clinical efficacy or safety are not a primary objective of the study.

DETAILED DESCRIPTION:
The main objective of the present proposal study is to assess the biological consequences of PARP inhibition in type I primary EC, in patients who receive therapy with AZD2281 during the period of time between diagnosis and surgery.

This is a phase 0 trial or "Exploratory Investigational New Drug" study, a type of trial that involves limited number of patient under drug therapy and has no therapeutic or diagnostic intent because the drug exposure has a limited duration and the dosage is lower than 100% of the dose required to yield a pharmacologic effect.

The purpose of the phase 0 studies is to assist in the go versus no-go decision-making process of a drug's fate earlier in the development process, using relevant human models instead of relying on sometimes inconsistent animal data, thus helping to confirm endpoints such as mechanism of action, pharmacology, bioavailability and pharmacodynamics.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically-confirmed type I primary endometrial carcinoma (EC). Diagnosis biopsy must contain 3-12 mg of tumour cellularity/stroma (Tumour: 5-20 mm) and this will be checked in the central laboratory for this trial. If tumour cellularity/stroma is inadequate, one re-biopsy with adequate tumour cellularity/stroma will be mandatory before study entry.
* WHO performance status ≤ 2.
* Adequate bone marrow function as shown by: ANC ≥ 1.5 x 109/L, Platelets ≥ 100 x 109/L, Hb >10g/dL.
* Adequate liver function as shown by:

serum bilirubin ≤ 1.5 x ULN INR < 1.3 (or < 3 on anticoagulants) ALT and AST ≤ 2.5x ULN

* Adequate renal function: serum creatinine ≤ 1.5 x mg/dL.
* Fasting serum cholesterol ≤300 mg/dL or ≤7.75 mmol/L and fasting triglycerides ≤ 2.5 x ULN.
* Signed informed consent, including consent to tissue collection and blood samples as specified by the protocol.

Exclusion Criteria:

* Subjects who have received prior anticancer therapies for the current endometrial cancer (including chemotherapy, radiotherapy, antibody based therapy, hormonotherapy or surgery).
* Patients, who have had a major surgery or significant traumatic injury within 4 weeks of start of study drug, patients who have not recovered from the side effects of any major surgery (defined as requiring general anesthesia) or patients that may require major surgery during the course of the study.
* Prior treatment with any investigational drug within the preceding 4 weeks.
* Patients receiving chronic, systemic treatment with corticosteroids or another immunosuppressive agent, except corticosteroids with a daily dosage equivalent to prednisone ≤ 20 mg. However, patients receiving corticosteroids must have been on a stable dosage regimen for a minimum of 4 weeks prior the study entry. Topical or inhaled corticosteroids are allowed.
* Patients who have received immunization with attenuated live vaccines within one week of study entry (note: during study period these kind of vaccines are also not allowed).
* Patients who have any severe and/or uncontrolled medical conditions or other conditions that could affect their participation in the study such as:

Symptomatic congestive heart failure of New York heart Association Class III or IV Unstable angina pectoris, myocardial infarction within 6 months of start of study drug, Serious uncontrolled cardiac arrhythmia or any other clinically significant cardiac disease Severely impaired lung function Uncontrolled diabetes as defined by fasting serum glucose >1.5 x ULN Active (acute or chronic) or uncontrolled severe infections Liver disease such as cirrhosis, chronic active hepatitis or chronic persistent hepatitis A known history of HIV seropositivity.

* Patients with an active, bleeding diathesis.
* Female patients who are pregnant or breast feeding, or adults of reproductive potential who are not using effective birth control methods. If barrier contraceptives are being used, these must be continued throughout the trial by both sexes. Hormonal contraceptives are acceptable as a sole method of contraception. (Women of childbearing potential must have a negative urine or serum pregnancy test within 7 days prior to administration of AZD2281).
* History of noncompliance to medical regimens.
* Patients unwilling to or unable to comply with the protocol.

Ages: 18 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patinets diagnosed with endometrial carcinoma prior surgery
Sampling Method: Non-Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2016-02; Primary Completion 2018-07 (Actual); Study Completion 2019-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Llombart, MD, PhD, Study Chair — Medica SIR
Locations (9):
- Spain (9):
  - MedSIR investigative site, A Coruña
  - MedSIR investigative site, Barcelona
  - MedSIR investigative site, Córdoba
  - MedSIR investigative site, Granollers
  - MedSIR, Madrid
  - MedSIR investigative site, Madrid
  - MedSIR investigative site, Santiago de Compostela
  - MedSIR investigative site, Valencia
  - MedSIR investigative site, Vigo

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Out of 49 patients initially considered for study eligibility, 9 did not sign the ICF and 4 did not meet eligibility criteria (screen failures).
  Out of 36 patients who were treated and included in the overall analysis and safety, 5 were excluded from the primary and secondary analysis because of no valid samples for biomarker characterization.
Period: Overall Study
Arm/Group | Olaparib
Started | 36
Samples Availability | 31 (31 of 36 patients had valid samples for analysis of biomarkers (primary and secondary analysis))
Completed | 33
Not Completed | 3
Not completed — Adverse Event | 3

BASELINE CHARACTERISTICS:
Population: A total of 36 patients were treated and included in the overall population and safety analyses.
Arm/Group | Olaparib
Number analyzed (Participants) | 36
Age, Categorical [Count of Participants; unit: Participants] — Population: 13 Screening Failures
  Participants
    <=18 years | 0
    Between 18 and 65 years | 19
    >=65 years | 17
Sex: Female, Male [Count of Participants; unit: Participants] — Population: 13 Screening Failures
  Participants
    Female | 36
    Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 35
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants] — Population: 13 Screening Failures
  participants
    Spain | 36

OUTCOME MEASURES:

1. Primary Outcome: Expression of Cell Cycle-related Proteins
Description: We assessed the change from baseline in the histological score (H-score) of the cell cycle-related proteins on endometrial tumor tissues after 28 (+/- 5) days of olaparib-based therapy. In detail, expression of the cyclin D1, Ki67, and caspase-3 active proteins evaluated by an H-score according to the following formula:
  H-score= 1x(%light staining) + 2x(%moderate staining) + 3x(%strong staining).
  The final score ranges from 0 to 300, where 0 indicates absence of staining (corresponding to the lowest tumor proliferation rate and better outcome) and 300 the maximum staining (corresponding to the highest tumor proliferation score and worse outcome).
Time Frame: Baseline and Day 28 (+/- 5)
Population: The analysis was performed in the complete population of analysis (N = 36) and in the population of biomarkers (N = 31).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Olaparib
Number analyzed (Participants) | 31
score on a scale
  Cyclin D1 pre-treatment - post-treatment | 46.1 (62.9)
  Ki67 pre-treatment - post-treatment | 0.8 (16.8)
  Caspase-3 active pre-treatment - post-treatment | 0.7 (9)
Statistical Analysis 1: Comparison: Olaparib; After having analyzed the H-score for each of 3 biomarkers, we calculated the change from baseline subtracting post-treatment H-score from baseline H-score. Data were expressed as mean value and relative standard deviation; Test type: Other — The P-valor Wilcoxon method is a non-parametric statistical hypothesis test used to evaluate changes from baseline H-score values of the three biomarkers; p = 0.033, Wilcoxon (Mann-Whitney) — In order to adjust the multiple comparisons made, Benjamini-Hochberg's false discovery rate (FDR) 10% method was used

2. Secondary Outcome: Protein Expression of Biomarkers Related to PARP-inhibition
Description: We assessed the change from baseline in the H-score of several biomarkers targeted by olaparib-based therapy on endometrial tumor tissues after 28 (+/- 5) days of treatment. In detail, expression of protein involved in the DNA repair (PARP1, ɣH2AX), angiogenesis (VEG, HIF-1α, PTEN), apoptosis (p65, p50, p53), glucose metabolism (GLUT1), proliferation (PH3), and regulation of gene transcription (ARID1A) were evaluated by an H-score according to the following formula:
  H-score= 1x(%light staining) + 2x(%moderate staining) + 3x(%strong staining).
  The final score ranges from 0 to 300, where 0 indicates absence of staining and 300 the maximum staining.
Time Frame: Baseline and Day 28 (+/- 5)
Population: The analysis was performed in the complete population of analysis (N = 36) and in the population of biomarkers (N = 31).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Olaparib
Number analyzed (Participants) | 31
score on a scale
  PARP1 pre-treatment - post-treatment | 10.3 (46.8)
  y-H2AX pre-treatment - post-treatment | -46.21 (67.7)
  VEGF pre-treatment - post-treatment | -9.4 (19.4)
  HIF-1α pre-treatment - post-treatment | 76.9 (74.3)
  PTEN pre-treatment - post-treatment | 3.2 (1)
  P65 pre-treatment - post-treatment | -0.2 (0.9)
  P50 pre-treatment - post-treatment | 0.1 (0.8)
  P53 pre-treatment - post-treatment | 0.1 (0.5)
  GLUT1 active pre-treatment - post-treatment | -20.8 (66.2)
  PHH3 pre-treatment - post-treatment | 3.1 (5.2)
  ARID1A pre-treatment - post-treatment | 20 (11)
Statistical Analysis 1: Comparison: Olaparib; After having analyzed the H-score for each of several biomarkers, we calculated the change from baseline subtracting post-treatment H-score from baseline H-score. Data were expressed as mean value and relative standard deviation; Test type: Other — The differences in the change from baseline of different biomarkers were evaluated by the P-valor Wilcoxon method, a non-parametric statistical hypothesis test; p = 0.03, Wilcoxon (Mann-Whitney) — In order to adjust the multiple comparisons made, Benjamini-Hochberg's false discovery rate (FDR) 10% method was used

3. Secondary Outcome: Plasma Levels of Olaparib
Description: Plasma concentration of olaparib administered at dosis of 300mg twice in a day (600mg/day). Values of plasma level of olaparib on days 7,14,21 and 28 were collected at time when maximum of drug concentration is reached. Data are reported as µg/mL.
Time Frame: Days 7,14,21 and 28
Population: The analysis was performed in the overall population of analysis (N = 36)
Measure: Mean (Standard Deviation); unit: µg/mL
Arm/Group | Olaparib
Number analyzed (Participants) | 36
µg/mL
  Day 07 | 6.55 (2.75)
  Day 14 | 5.61 (2.7)
  Day 21 | 6.49 (2.95)
  Day 28 | 4.7 (3.13)

4. Secondary Outcome: Number of Participants With Olaparib-Associated Toxicities
Description: To assess the tolerability for all treated patients (N=36) according to NCI-CTCAE v.4.03.
Time Frame: Up to 28 days (+/- 5)
Population: The analysis was performed in the complete population of analysis (N = 36) and took in account patients who discontinued study for drug-associated toxicity.
Measure: Count of Participants; unit: Participants
Arm/Group | Olaparib
Number analyzed (Participants) | 36
Participants | 3

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the first day of treatment initiation until to 28 days (+/- 7 days) after the last day of study treatment.
Arm/Group | Olaparib
All-Cause Mortality (participants affected / at risk) | 0/36
Serious Adverse Events (participants affected / at risk) | 1/36
Other Adverse Events (participants affected / at risk) | 15/36
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Olaparib (N=36)
Post-surgical wound infection (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Olaparib (N=36)
Nausea (Gastrointestinal disorders) | 15
Neutropenia (Blood and lymphatic system disorders) | 10
Anemia (Blood and lymphatic system disorders) | 9
Asthenia (General disorders) | 9
Vomiting (Gastrointestinal disorders) | 6
Diarrhea (Gastrointestinal disorders) | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2016-11-03): https://cdn.clinicaltrials.gov/large-docs/16/NCT02506816/Prot_000.pdf
  • Statistical Analysis Plan (2017-12-11): https://cdn.clinicaltrials.gov/large-docs/16/NCT02506816/SAP_002.pdf